CLINICAL TRIAL: NCT03598712
Title: Interest of Local Compression by Thoracic Bandage on the Management of Seroma in Patients Treated by Mastectomy With or Without Lymphadenectomy. Local Compression Seroma DIminution Objective
Brief Title: Local Compression Seroma DIminution Objective (CLODIS)
Acronym: CLODIS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Surgical practices have evolved as surgeons practice immediate reconstructive surgery. We have not been able to meet the recruitment target.
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLODIS
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Mastectomy; Seroma
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Punctures

STUDY DESIGN:
Intervention Model Description: Phase 3 prospective, randomized, monocentric controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression by chest bandage urgo K2® (Experimental): After the second puncture, the local compression by thoracic bandage will be put in place.
  The system being effective 7 days, it will be left in place between each visit. A visit will be made for all patients 7 days after the installation of the device. However, if necessary, an intermediate visit may be carried out.
  During these visits, a puncture will be made according to the criteria mentioned above. The bandage will be renewed after each visit.
  The device will be removed after 15 days without indication of a new puncture. The patient will be seen again between 10 and 15 days after the bandage is removed for a final evaluation.
  Interventions: Device: Compression by chest bandage urgo K2®; Procedure: punctures
- punctures (Active Comparator): After the second puncture, the patient will be seen at the same frequency as in the experimental arm.
  The decision to perform a puncture will be made according to the same criteria and the follow-up conditions will be identical.
  Interventions: Procedure: punctures

INTERVENTIONS:
Device: Compression by chest bandage urgo K2® — 1. - Installation of a short stretch belt (urgo K2® kit)
  2. - Installation of a long stretch cohesive band providing additional pressure necessary to reach therapeutic pressure and maintain the device (urgo K2® kit).
  3. - Control of the pressure exerted by the bandage by the "KIKUHIME® Sub Bandge pressure Monitor" device
  Arms: Compression by chest bandage urgo K2®
Procedure: punctures — Every 7 days after the second puncture of a volume > 250ml of seroma, the patients are examined by 2 practitioners. They define the indication of the puncture. The seroma is aspirated after a skin puncture with a needle connected with a Redon® drain.

SUMMARY:
This study evaluates the impact of local compression by chest bandage on the number of seroma punctures in patients treated by mastectomy with or without lymphadectomy. Half of the participants will have local compression by chest bandage in addition to seroma punctures while the other half will only have punctures.

DETAILED DESCRIPTION:
The most common complication induced by mastectomy is seroma formation. This seroma is a serolymphatic effusion that is created in the days following surgery. Iterative puncture is the only treatment for seroma mentioned in the literature. A retrospective study in the investigator's establishment on 1800 patients determined that a second puncture greater than 250ml is predictive of a chronicisation of punctures. The research hypothesis is that by applying local compression by chest bandaging with the Urgo® K2 kit, the "dead space" created by surgery would be removed. This would help resorb the seroma and reduce the number of punctures.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for histologically proven breast cancer treated by total mastectomy, whether or not dissociated from the sentinel node technique, with or without axillary curing.
* Patient with a second seroma puncture with a volume greater than or equal to 250 ml.
* Neo adjuvant chemotherapy authorized.
* Absence of known metastases.
* Patient has given written consent.

Exclusion Criteria:

* Mastectomy with immediate reconstruction.
* Partial mastectomy.
* Concurrent bilateral mastectomy.
* Delay in healing observed at inclusion.
* Patient under legal protection.
* Chronic respiratory failure.
* Patient with a pacemaker.
* Personality disorders and known progressive psychiatric pathology.
* Inability to submit to trial follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Number of puncture(s) after inclusion in both patient groups | 180 days
  In each group, we will count the number of punctures performed after the 2nd puncture with a volume > 250ml (inclusion).

SECONDARY OUTCOMES:
The time required to take charge of adjuvant treatments | 180 days
  Deferral of adjuvant therapy related to seroma: Treatment regimen and adjuvant appointments will be collected at inclusion. Each deviation will be analyzed and attributed or not to the presence or complications of seroma.
Volume punctured after inclusion in both patient groups. | 180 days
  For each new puncture, the volume of serolymphatic fluid will be measured and the time between two punctures analyzed
comparison of the average change Quality of life scores between each arm | 180 days
  Quality of life is assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, for the cancer in general and EORTC QLQ-BR23 specifically for the breast cancer (study inclusion and exit). The EORTC QLQ-C30 questionnaire, resulting in a score for the quality of life between 0 to 100.
comparison of the average change anxiety scores between each arm | 180 days
  Anxiety / depressions are assessed by the Hospital Anxiety and Depression scale (study inclusion and exit)
comparison of the average change Pain scores between each arm | 180 days
  1. Numerical rating scale for pain (EN) The EN evaluates levels of pain intensity using an 10-point scale (range 0-10), with 0 being classified as "no sensation", 3 "pain threshold", 10 "pain as bad as could be.(at each visit),
  2. Neuropathic Pain (DN4) (inclusion and study exit)
The aesthetic impact on the puncture site. | 180 days
  The evaluation of the aesthetic impact on the puncture zone will be carried out by comparing the photographs taken at the inclusion, during the visit to the consultation at 10-15 days after the last puncture (for the standard arm) and at 10-15 days after the removal of the bandage device and finally during the consultation with the oncologist.
Validation of a score allowing the description of the seroma of grades 2 and the indication of a puncture | 180 days
  Based on the observation grids carried out by the 2 professionals during a separate evaluation, we compare the 4 items defined to the indication chosen for the puncture as well as the volume of puncture when it is carried out.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - TANQUEREL Julie, Caen
  - Centre Françis Baclesse, Caen

IPD SHARING:
Plan to Share IPD: No